CLINICAL TRIAL: NCT00249405
Title: Predicting Alcoholics' Treatment Responses to an SSRI
Brief Title: Predicting Alcoholics' Treatment Responses to a Selective Serotonin Re-uptake Inhibitor (SSRI)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Robert Anthenelli, M.D., Principle Investigator
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NIAAAANT013957-B; R01AA013957 (NIH); NIH Grant R01 AA013957-02
Record Dates: First submitted 2005-11-04; First posted 2005-11-07 (Estimated); Last update posted 2010-11-03 (Estimated); Status verified 2010-11

CONDITIONS: Alcoholism; Alcohol Abuse
Keywords: Clinical trial; Alcoholism; Alcohol; Pharmacogenetics; Citalopram; Genotype; Therapy compliance; Serotonin inhibitor; Alcoholism/alcohol abuse therapy
MeSH Terms: conditions — Alcoholism; Patient Compliance | interventions — Citalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): citalopram
  Interventions: Drug: Citalopram + MI
- 2 (Placebo Comparator): Placebo
  Interventions: Behavioral: Placebo + MI

INTERVENTIONS:
Drug: Citalopram + MI — 14-week citalopram treatment + Motivational Interview (MI) and 9 brief sessions of a manual-guided Compliance Enhancement Therapy; post-treatment follow-up assessments will be conducted at 4, 12 and 24 weeks.
  Other Names: celexa
  Arms: 1
Behavioral: Placebo + MI — placebo + single Motivational Interview (MI) and 9 brief sessions of a manual-guided Compliance Enhancement Therapy; post-treatment follow-up assessments will be conducted at 4, 12 and 24 weeks.
  Arms: 2

SUMMARY:
This study is being done to determine if citalopram is safe and effective in the treatment of alcohol dependence. A second purpose is to evaluate whether alcohol dependent individuals who differ in a specific genetic marker respond differently to citalopram.

Citalopram is a drug approved by the U.S. Food and Drug Administration (FDA) for the treatment of depression. It belongs to a category of medications called selective serotonin re-uptake inhibitors or SSRIs. The U.S. FDA has not approved citalopram for the treatment of alcohol dependence. Therefore, it is being used "off-label" in this study.

DETAILED DESCRIPTION:
Relapse to alcoholism remains a vexing clinical and national health problem. Efforts to match alcohol dependent patients to specific treatments based on their clinical characteristics have produced mixed results. Pharmacogenetics (the study of genetic influences on therapeutic response to drugs) offers a powerful new tool to match specific elements of an individual patient's complex genetic blueprint with targeted pharmacotherapies to which that individual may optimally respond.

The purpose of this proposed research is to apply pharmacogenetic techniques to predict which alcohol dependent patients will respond favorably to a trial of a selective serotonin re-uptake inhibitor (SSRI) for the prevention of alcoholism relapse. Our central hypothesis is that genetic differences affecting serotonin transporter function will influence an alcohol dependent individual's treatment response to the SSRI, citalopram. To test this hypothesis, we will perform a 14-week, randomized, double blind, parallel group comparison of citalopram and placebo in treatment seeking outpatients who meet DSM-IV criteria for alcohol dependence. All subjects will receive a single Motivational Interview and 9 brief sessions of a manual-guided Compliance Enhancement Therapy designed to promote treatment adherence and enhance motivation to quit or cut down on drinking. Post-treatment follow-up assessments will be conducted at 4, 12 and 24 weeks. Subjects' DNA will be genotyped to determine allelic variants in the promoter region of the serotonin transporter gene that have been found to markedly affect serotonin reuptake and influence treatment responsiveness to SSRIs.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with a diagnosis of DSM-IV alcohol dependence
* Not morbidly obese or underweight
* Express desire to quit or cut down on drinking for duration of trial

Exclusion Criteria:

* Clinically significant laboratory evidence of diseases
* Have active psychological disorders other than alcoholism

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2005-02; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Percent days abstinent | 24 weeks

SECONDARY OUTCOMES:
Percent heavy drinking days | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert M. Anthenelli, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Thompson RD, Heffner JL, Strong JA, Blom TJ, Anthenelli RM. Relationship between the serotonin transporter polymorphism and obsessive-compulsive alcohol craving in alcohol-dependent adults: a pilot study. Alcohol. 2010 Aug;44(5):401-6. doi: 10.1016/j.alcohol.2010.05.008. Epub 2010 Jul 3. PMID 20598843
- [Derived] Heffner JL, Tran GQ, Johnson CS, Barrett SW, Blom TJ, Thompson RD, Anthenelli RM. Combining motivational interviewing with compliance enhancement therapy (MI-CET): development and preliminary evaluation of a new, manual-guided psychosocial adjunct to alcohol-dependence pharmacotherapy. J Stud Alcohol Drugs. 2010 Jan;71(1):61-70. doi: 10.15288/jsad.2010.71.61. PMID 20105415